CLINICAL TRIAL: NCT01571479
Title: The Feasibility and Safety of a Three-Port Laparoscopic Cholecystectomy Using a 2-mm Mini-Instrument
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Kwan Woo Kim, Haeundae paik hospital, Inje University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-026
Record Dates: First submitted 2012-03-31; First posted 2012-04-05 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Gallbladder Disease
Keywords: laparoscopic cholecystectomy; mini-instrument
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2-mm mini-instrument (M-LC) (No Intervention): M-LC is three-port laparoscopic cholecystectomy using a 2-mm mini-instrument.
  Interventions: Procedure: 2- mini-instrument
- conventional instrument(C-LC) (No Intervention): C-LC is conventional three port laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: 2- mini-instrument — The patient was positioned in the supine position with the head and right side up.
  Under general anesthesia, pneumoperitoneum (12 mmHg) was established after an 11-mm port was placed through 11-mm transumbilical incision by the open method.
  A 10-mm 0-degree laparoscope was inserted through this umbilical port. A 5-mm trocar was then placed in the epigastric area, and the surgeon determined through 'laparoscopic surgical view' whether the 2-mm mini-instrument could be used as the right subcostal port . If the 2-mm mini-instrument could be used as the right subcostal port, a 2-mm trocar was inserted . If not, a 5-mm trocar was inserted for the right subcostal port. Therefore, this point is the unique difference between the two groups.
  Other Names: micro-instrument
  Arms: 2-mm mini-instrument (M-LC)

SUMMARY:
The aim of this study was to show that this technique is feasible, safe and easily reproducible and to evaluate the selection criteria for a three-port laparoscopic cholecystectomy using a 2-mm mini-port.

DETAILED DESCRIPTION:
Since the first four-port laparoscopic cholecystectomy (LC) was reported in 1987, various surgical options for LC have been developed. Recently, single port LC (SPLC) has been increasingly performed to minimize tissue trauma, improve cosmesis and decrease postoperative pain for patients. Some surgeons suggest that the four- or three-port LC using mini-ports could be as safe, effective, economical and cosmetic as SPLC. For this reason, the investigators started M-LC for patients with benign gallbladder disease in April 2010.

Prospectively collected data from 133 patients who underwent LC for benign gallbladder disease between April 2010 and April 2011 were retrospectively reviewed.

The patient's selection for M-LC was determined by surgeon's judgment based on 'laparoscopic surgical view' after inserting the laparoscope in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* all patients required laparoscopic cholecystectomy for benign gallbladder diseases.

Exclusion Criteria:

* open cholecystectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with complications or open conversion to M-LC | one year

CONTACTS AND LOCATIONS:
Overall Officials: kwan woo kim, Principal Investigator — University of Inje College of Medicine, Haeundae Paik Hopsital
Locations (1):
- University of Inje College of Medicine, Haeundae Paik Hopsital, Busan, South Korea

REFERENCES:
- [Result] Aprea G, Coppola Bottazzi E, Guida F, Masone S, Persico G. Laparoendoscopic single site (LESS) versus classic video-laparoscopic cholecystectomy: a randomized prospective study. J Surg Res. 2011 Apr;166(2):e109-12. doi: 10.1016/j.jss.2010.11.885. Epub 2010 Dec 22. PMID 21227454
- [Result] Bisgaard T, Klarskov B, Trap R, Kehlet H, Rosenberg J. Microlaparoscopic vs conventional laparoscopic cholecystectomy: a prospective randomized double-blind trial. Surg Endosc. 2002 Mar;16(3):458-64. doi: 10.1007/s00464-001-9026-5. Epub 2001 Nov 16. PMID 11928028
- [Result] Chow A, Purkayastha S, Aziz O, Pefanis D, Paraskeva P. Single-incision laparoscopic surgery for cholecystectomy: a retrospective comparison with 4-port laparoscopic cholecystectomy. Arch Surg. 2010 Dec;145(12):1187-91. doi: 10.1001/archsurg.2010.267. PMID 21173293
- [Result] Curcillo PG 2nd, Wu AS, Podolsky ER, Graybeal C, Katkhouda N, Saenz A, Dunham R, Fendley S, Neff M, Copper C, Bessler M, Gumbs AA, Norton M, Iannelli A, Mason R, Moazzez A, Cohen L, Mouhlas A, Poor A. Single-port-access (SPA) cholecystectomy: a multi-institutional report of the first 297 cases. Surg Endosc. 2010 Aug;24(8):1854-60. doi: 10.1007/s00464-009-0856-x. Epub 2010 Feb 5. PMID 20135180
- [Result] Edwards C, Bradshaw A, Ahearne P, Dematos P, Humble T, Johnson R, Mauterer D, Soosaar P. Single-incision laparoscopic cholecystectomy is feasible: initial experience with 80 cases. Surg Endosc. 2010 Sep;24(9):2241-7. doi: 10.1007/s00464-010-0943-z. Epub 2010 Mar 3. PMID 20198490
- [Result] Elsey JK, Feliciano DV. Initial experience with single-incision laparoscopic cholecystectomy. J Am Coll Surg. 2010 May;210(5):620-4, 624-6. doi: 10.1016/j.jamcollsurg.2009.12.030. PMID 20421017
- [Result] Franklin ME Jr, Jaramillo EJ, Glass JL, Trevino JM, Berghoff KR. Needlescopic cholecystectomy: lessons learned in 10 years of experience. JSLS. 2006 Jan-Mar;10(1):43-6. PMID 16709356
- [Result] Gagner M, Garcia-Ruiz A. Technical aspects of minimally invasive abdominal surgery performed with needlescopic instruments. Surg Laparosc Endosc. 1998 Jun;8(3):171-9. PMID 9649038